CLINICAL TRIAL: NCT04304573
Title: Is Correcting Total Serum Calcium Levels for Serum Albumin Necessary in Assessing Symptomatic Hypocalcemia After Total Thyroidectomy: a Prospective Cohort Study
Brief Title: Is Correcting Total Serum Calcium Levels Important After Thyroidectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Andro Košec, MD, PhD, Consultant Otorhinolaryngologist and Head and Neck Surgeon, University Hospital
Other Study IDs: KBCSM13
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Hypocalcemia; Thyroid; Parathyroid Dysfunction; Calcium Disorder; Hormone Disturbance; Postoperative Complications
Keywords: hypocalcemia; total thyroidectomy; Payne's formula; ionized calcium; parathyroid hormone; predictive factor
MeSH Terms: conditions — Hypocalcemia; Thyroid Diseases; Parathyroid Diseases; Endocrine System Diseases; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with hypocalcemia symptoms and low serum calcium: Patients with postoperative hypocalcemia defined as serum calcium levels < 2.00 mmol/L. Patients may have low or normal PTH range (defined by the Department of Laboratory Diagnostics reference range from 1.6 to 6.9 pmol/L)
  Interventions: Diagnostic Test: Total serum calcium blood test
- Patients with hypocalcemia symptoms and normal serum calcium: Patients with hypocalcemia symptoms but without postoperative hypocalcemia defined as serum calcium levels > 2.00 mmol/L. Patients may have low or normal PTH range (defined by the Department of Laboratory Diagnostics reference range from 1.6 to 6.9 pmol/L)
  Interventions: Diagnostic Test: Total serum calcium blood test

INTERVENTIONS:
Diagnostic Test: Total serum calcium blood test — Total serum calcium measurements will be done on the first postoperative day. Also ionized calcium, corrected total serum calcium for serum albumin with Payne's formula and PTH will be monitored.

SUMMARY:
This study is designed as a prospective non-randomized longitudinal single- center cohort study to evaluate the importance of correcting total serum calcium levels. It will enroll around 100 patients undergoing total thyroidectomy with data being collected from March 2020 up to August 2020. The aim of this study is to determine whether total serum calcium level should be corrected for serum albumin in assessing symptomatic hypocalcemia after total thyroidectomy and which variable (total serum calcium, ionized calcium, corrected serum calcium for albumin with Payne's formula or early PTH) is the most valuable predictor of symptomatic hypocalcemia after total thyroidectomy.

DETAILED DESCRIPTION:
This study is designed as a prospective non-randomized longitudinal single- center cohort study to evaluate the importance of correcting total serum calcium levels. It will enroll around 100 patients undergoing total thyroidectomy with data being collected from March 2020 up to August 2020.The patients will be eligible if they undergo total thyroidectomy regardless of the surgical indication, if complete serum PTH and calcium data are available through the first five postoperative days and if they sign an informed consent form. Patients with incomplete data, preoperative pathological calcium or PTH levels, or suffering from conditions affecting calcium metabolism and parathyroid function will be excluded from the study.

Demographic and clinical data including age, sex, preoperative and postoperative laboratory values (total serum calcium, ionized calcium, corrected total serum calcium for serum albumin and PTH), neck dissection procedures, and postoperative calcium supplement therapy will be noted.

Primary outcome measures are presence of hypocalcemia on the first and fifth postoperative day. Secondary outcome measures are the need for calcium supplement therapy during the first five postoperative days, amount of medication given and correlation between presence of symptoms and low values of corrected total serum calcium levels. Preoperative blood samples for serum PTH and calcium measurements will be obtained after hospital admission. Postoperative serum PTH will be sampled 1 hour after surgery and at 7 am on the firstand fifth postoperative day. Serum calcium sampling will be performed daily if a patient has hypocalcemia detected on the first postoperative day. Hypocalcemia is defined as serum calcium levels < 2.00 mmol/L regardless of clinical symptoms present. Normal PTH range is defined by the Department of Laboratory Diagnostics reference range - from 1.6 to 6.9 pmol/L. The recovery of parathyroid function is defined as the return of serum PTH and serum calcium to normal values, requiring no further calcium or vitamin D supplementation. If the patient does not have laboratory or clinical signs of hypocalcemia, calcium supplement therapy will not be administered. Supplement therapy will be administered in patients with laboratory findings confirming hypocalcemia. Supplement therapy consists of either peroral elemental calcium (calcium carbonate, 1-gram unit) or calcitriol (0.5 microgram unit) or both. If postoperative calcium and PTH are normal and there are no symptoms of discomfort, the patient will be discharged on the first or second postoperative day and serum PTH and calcium sampling will be performed on an outpatient basis. If the patient did not receive treatment during hospitalization, no supplements will be prescribed after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* The patients were eligible if they underwent total thyroidectomy regardless of the surgical indication, if complete serum PTH and calcium data were available through the first five postoperative days and if they signed an informed consent form.

Exclusion Criteria:

* Patients with incomplete data, preoperative pathological calcium or PTH levels, or suffering from conditions affecting calcium metabolism and parathyroid function were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total thyroidectomy regardless of the surgical indication.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-09 (Estimated); Primary Completion 2020-08-09 (Estimated); Study Completion 2020-09-09 (Estimated)

PRIMARY OUTCOMES:
Corrected total serum calcium value | 5 days
  Statistically significant correlation between low value of corrected total serum calcium level for albumin and hypocalcemia symptoms

SECONDARY OUTCOMES:
Administration of postoperative calcium supplement therapy | 5 days
  Whether or not, and the amount of postoperative calcium supplement therapy needed in case of hypocalcemia.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Rašić, MD,PhD, Study Chair — Department of Otorhinolaryngology and Head and Neck Surgery
Locations (1):
- University Hospital Center Sestre milosrdnice, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No